CLINICAL TRIAL: NCT02969395
Title: Pacing Capture Threshold Change Following 3T MRI Scan of MR Conditional Cardiac Implantable Electronic Devices
Brief Title: 3T MRI CIED Post-Approval Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 3T
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Rhythm Disorder
Keywords: 3T; Magnetic Resonance Imaging (MRI); Implantable Cardioverter Defibrillator (ICD); Implantable Pulse Generator (IPG); Cardiac Resynchronization Therapy (CRT); Cardiac Implantable Electronic Device (CIED)
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate product performance of Magnetic Resonance (MR) Conditional Cardiac Implantable Electronic Devices (CIED) following 3 tesla (3T) MRI exposure. This will be achieved by evaluating the changes in pacing capture threshold (PCT) measurements following 3T MRI scan exposure. This study is required by FDA as a condition of approval of 3T MRI compatible labeling of applicable CIED systems. This study is conducted within Medtronic's post-market surveillance platform, the Product Surveillance Registry (PSR).

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Subject is intended to be implanted or is within 30 days post-implant of a qualifying Medtronic 3T MR Conditional CIED system

Exclusion Criteria:

* Subject who is, or will be inaccessible for follow-up at a study site
* Subject with exclusion criteria required by local law (Europe, Central Asia [ECA] only)
* Implant and follow-up data, including any adverse device effects and system modifications at implant through the time of enrollment are unavailable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients intended to be implanted or are within 30 days post-implant of a qualifying Medtronic 3T MR Conditional CIED system. All subjects must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-04; Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
The proportion of patients implanted with an MR Conditional CIED System with a pre-MRI to post-MRI scan PCT measure change of >0.5 Volts following 3T MRI scan exposure. | Patients will be followed for approximately 5 years.

CONTACTS AND LOCATIONS:
Locations (204):
- United States (118):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Chandler, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - La Quinta, California
  - Los Angeles, California
  - Palm Springs, California
  - Rancho Mirage, California
  - Redwood City, California
  - Salinas, California
  - San Diego, California
  - San Francisco, California
  - Stanford, California
  - Torrance, California
  - Van Nuys, California
  - Centennial, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Davenport, Florida
  - Davie, Florida
  - Jacksonville, Florida
  - Panama City, Florida
  - Safety Harbor, Florida
  - Sebastian, Florida
  - Tampa, Florida
  - Albany, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Clinton, Maryland
  - Hyattsville, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Lansing, Michigan
  - Marquette, Michigan
  - Ypsilanti, Michigan
  - Coon Rapids, Minnesota
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - Hattiesburg, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Eatontown, New Jersey
  - Morristown, New Jersey
  - Ocean Township, New Jersey
  - Ridgewood, New Jersey
  - Albuquerque, New Mexico
  - Bay Shore, New York
  - Garden City, New York
  - Huntington, New York
  - Manhasset, New York
  - New Hyde Park, New York
  - New York, New York
  - Poughkeepsie, New York
  - Staten Island, New York
  - Suffern, New York
  - The Bronx, New York
  - Utica, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Tyler, Texas
  - Burlington, Vermont
  - Arlington, Virginia
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (5):
  - Brussels
  - Dinant
  - Leuven
  - Liège
  - Yvoir
- Canada (6):
  - Kingston, Ontario
  - Sainte-Foy, Quebec
  - Calgary
  - Montreal
  - Ottawa
  - Trois-Rivières
- China (3):
  - Kunming
  - Taiyuan
  - Tianjin
- Copenhagen, Denmark
- France (11):
  - Avignon
  - Brest
  - Clermont-Ferrand
  - Dijon
  - La Rochelle
  - Metz-Tessy
  - Montpellier
  - Nantes
  - Paris
  - Pringy
  - Saint-Priest-en-Jarez
- Germany (7):
  - Aachen
  - Cologne
  - Essen
  - Hanover
  - Homburg
  - Tübingen
  - Ulm
- Athens, Greece
- Budapest, Hungary
- Italy (4):
  - Castrovillari
  - Lecce
  - Milan
  - Udine
- Japan (11):
  - Fuchū
  - Hidaka
  - Hirosaki
  - Hiroshima
  - Kawasaki
  - Kitakyushu
  - Kyoto
  - Ōsaka-sayama
  - Sapporo
  - Toyoake
  - Urasoe
- Kuala Lumpur, Malaysia
- Netherlands (4):
  - Eindhoven
  - Maastricht
  - Nieuwegein
  - Rotterdam
- Creixomil, Portugal
- Belgrade, Serbia
- Košice, Slovakia
- Ljubljana, Slovenia
- South Korea (9):
  - Busan
  - Changwon
  - Daegu
  - Gangneung
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Seongnam-si
  - Seoul
- Spain (9):
  - A Coruña
  - Granada
  - Madrid
  - Palma de Mallorca
  - Salamanca
  - Santa Cruz de Tenerife
  - Santiago de Compostela
  - Valencia
  - Valladolid
- Skövde, Sweden
- Switzerland (3):
  - Geneva
  - Lausanne
  - Zurich
- United Kingdom (5):
  - Birmingham
  - Leicester
  - Liverpool
  - Manchester
  - Middlesbrough